CLINICAL TRIAL: NCT00395590
Title: A Cross Sectional Study of Patients With Obstructive Sleep Apnea for Polymorphisms in Genes of Inflammatory Cytokines.
Brief Title: Polymorphisms in Inflammatory Cytokines Genes in Subjects With Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Other Study IDs: 5594ctil
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Last update posted 2006-11-03 (Estimated); Status verified 2005-02

CONDITIONS: Sleep Apnea
Keywords: OSA inflammatory cytokines, metabolic syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Obstructive sleep apnea is a common sleep disorder. It is known to be related with increased body mass, abdominal obesity, insulin resistance and hypertension. It is currently believed to be a feature of the metabolic syndrome. Other features of the metabolic syndrome-such as insulin resistace were found related to inflammation and inflammatory cytokines. Several polymorphisms in the genes that encode interleukin 6,inteleukin 10 and TNF-alpha have significant influence on the amounts of cytokine production. we thus hypothesize that polymorphisms related to increased pruduction are more common in subjects with OSA than in matched controls

DETAILED DESCRIPTION:
Patients attending a sleep apnea clinic for evluation will be recruited. Patients found positive for OSA will be compared to the patients with a negative study for OSA for the prevalence of polymorphisms in genes of inflammatory cytokines and cytokine levels

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the sleep apnea clinic for evaluation

Exclusion Criteria:

* patients known to have inflammatory conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-11; Study Completion 2007-11

CONTACTS AND LOCATIONS:
Overall Officials: mates mates, MD, Study Director — Ben-Gurion University of the Negev